CLINICAL TRIAL: NCT03569163
Title: Accuracy of Pulse Oximeters With Profound Hypoxia
Brief Title: Pulse Oximeter Test
Status: Completed | Type: Observational
Sponsor: Spry Health (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: SpryHealth
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Spry Loop oximeter — Oximetry was performed on the subjects and accuracy was determined based on comparison with blood gas analysis.

SUMMARY:
Assessment of Spry Health's Loop oximetry accuracy in profound hypoxia

ELIGIBILITY:
Inclusion Criteria:

* Good general health with no evidence of medical problems

Exclusion Criteria:

* Smoking
* Anemia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 11 healthy adults
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Oximetry Accuracy | 30 minutes
  RMSE of pulse oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Hypoxia Lab, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No